CLINICAL TRIAL: NCT00479115
Title: AMD3100 in Combination With G-CSF to Mobilize Peripheral Blood Stem Cells in Patients With Fanconi Anemia(FA): A Phase I/II Study
Brief Title: Mobilization and Collection of Peripheral Blood Stem Cells in Patients With Fanconi Anemia Using G-CSF and AMD3100
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CCHMCEH004; R01HL081499 (NIH)
Record Dates: First submitted 2007-05-23; First posted 2007-05-25 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Fanconi Anemia
MeSH Terms: conditions — Fanconi Anemia | interventions — plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMD3100 (Experimental)
  Interventions: Drug: AMD3100; Device: AmCell CliniMACs

INTERVENTIONS:
Drug: AMD3100 — 240 mcg/kg subcutaneously, minimum of two days; maximum of eight days
Device: AmCell CliniMACs — CD34+ cell selection from peripheral collection

SUMMARY:
The purpose of this research study is to determine whether an experimental drug called AMD3100 used in combination with another medication called G-CSF is safe and can help to increase the amount of blood stem cells (called CD34+ stem cells) found in the peripheral blood of patients with Fanconi anemia. While AMD3100 has been used successfully in adult volunteers and cancer patients, it has not been used in children or patients with Fanconi anemia and in only a few children with cancer.

Fanconi anemia is a rare genetic disease. Most Fanconi anemia patients eventually develop bone marrow failure, a condition in which the bone marrow no longer produces red blood cells (to carry oxygen), white blood cells (to fight infection), and platelets (to help blood clot). The only successful treatment for patients with Fanconi anemia with bone marrow failure is bone marrow transplantation. However, this treatment has many risks and is not available to all patients with Fanconi anemia.

CD34+ cells include stem cells found in the bone marrow or peripheral blood which are capable of making the red blood cells, white blood cells, and platelets. CD34+ stem cells can be collected from bone marrow or peripheral blood and purified using an experimental device called the CliniMACS. However, most Fanconi anemia patients do not have enough CD34+ stem cells in their bone marrow or peripheral blood to be collected using standard methods that work well in children and adults who don't have Fanconi anemia.

DETAILED DESCRIPTION:
Fanconi anemia is a rare autosomal recessive syndrome comprised of progressive bone marrow failure, congenital anomalies and a predisposition to malignancy. The heterozygote rate in the United States may be as high as 1 in 300. The mean age for the onset of aplastic anemia is approximately eight years. Although improved supportive care has prolonged the survival of these patients from only a few years from the diagnosis of bone marrow failure, the mean age of death is still approximately 24 years of age. Most patients die from complications of bone marrow failure including bleeding, or infection, or from malignancy or complications of stem cell transplantation. In a recent 20 year review of patients in the Fanconi anemia registry, the actual risk of developing leukemia or other cancers was approximately 30%.

The diagnosis of Fanconi anemia initially rested upon finding the combination of bone marrow failure with congenital anomalies. These anomalies include cafe au lait spots and/or hypo pigmentation of the skin, short stature, upper limb malformations (often involving the thumb or radius), renal and gastrointestinal abnormalities, microcephaly, and characteristic facies with a broad nasal base, epicanthal folds, narrow set and small eyes and micrognathia. The bone marrow failure is characterized by slow progression to severe bone marrow aplasia and pancytopenia, stress erythropoiesis with fetal features including macrocytosis, elevated hemoglobin F, and i antigen expression. Attempts to culture bone marrow progenitors in vitro from patients with Fanconi anemia demonstrates decreased numbers of myeloid and erythroid colonies (CFU) consistent with clinical bone marrow failure.

Fanconi anemia cells appear to have a defect in DNA repair that leads to increased spontaneous chromosomal breakage. This feature increases the susceptibility of Fanconi anemia cells to DNA bifunctional cross-linking agents such as mitomycin C and diepoxybutane (DEB). The diagnosis of Fanconi anemia now relies upon detecting increased chromosomal breakage after in vitro treatment with DEB. 11 Similarly, cells cultured from patients with Fanconi anemia display increased susceptibility to the cytotoxicity of mitomycin C. More recently, cells from patients with Fanconi anemia have been demonstrated to display G2 phase prolongation/arrest, increased sensitivity to toxicity by oxygen, defective p53 induction and increased apoptosis.

Fanconi anemia can be classified into at least thirteen complementation groups by somatic cell hybrids. The complementation is based upon correction of the chromosomal sensitivity to cross-linking agents in hybrid cells. Twelve independent genes have been cloned and characterized within these 13 complementation groups. A loss of function in any of these genes including FANC A, B, C, D2, E, F, G, J, L, M, N, and FANC D1 (which is BRCA2) can cause Fanconi anemia. However, complementation groups A, C, and G account for approximately 80-85% of patients with Fanconi anemia in the United States. Discrete mutations in these genes have been identified in families with the disorder. Expression of the complementary cDNA gene in the respective Fanconi anemia cells in vitro corrects the increased chromosomal breakage from DEB and the increased sensitivity to mitomycin C. Expression of gene products in bone marrow progenitors from patients with Fanconi anemia increases survival in in vitro assays.

The current treatment for Fanconi anemia relies upon hematological support in the form of red blood cell and platelet transfusions. Aplastic anemia will transiently respond to androgen therapy in 50% of children. G-CSF has also been utilized in published studies from our own group to improve the number of myeloid cells in the peripheral circulation. Bone marrow transplantation has cured some patients of their bone marrow failure; however, there appears to be more toxicity to the conditioning regimens and there may be increased numbers of solid tumors post transplant compared to patients without the disorder. Survival five years after a matched sibling transplant now exceeds 65% and after an unrelated donor transplant 30%. More recent studies in unrelated donor transplant for Fanconi anemia at Cincinnati Children's Hospital and the University of Minnesota have reported survival rates approaching those observed in matched sibling donor transplants. However, graft failure resulting in death remains a major obstacle. The availability of sufficient numbers of (previously purified and cryopreserved) autologous HSC for re-infusion after graft failure may prevent this complication.

Finally, gene therapy approaches are being pursued, but to date, there is no evidence for cure with this approach in humans, although correction has been reported in murine models. These studies are hampered by the fact that mouse knockouts of FA genes do not develop spontaneous aplastic anemia and thus are not phenocopies of the human disease. Thus in previously reported mouse-studies, gene therapy approaches required ablative total body irradiation of the recipient mice to ensure engraftment of the gene corrected stem cells.

An obvious limitation of Fanconi anemia hematopoietic stem cell gene transfer is that the necessary target for genetic manipulation, the hematopoietic stem cell (or its surrogate, CD34+ cell) is progressively lost during the development of aplastic anemia. Thus at the time of severe aplasia and the greatest need for treatment, target stem cells for genetic modification are deficient. Collection of a meaningful number of HSC prior to the onset of aplastic anemia for eventual use in a therapeutic gene therapy trial will be explored in the study outlined here. Key questions remaining are whether corrected HSC from Fanconi anemia patients will engraft after autologous re-infusion without any cyto-reductive treatment of the recipient and, if engrafted, whether the corrected cells will demonstrate a proliferative advantage over uncorrected stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have had a diagnosis of Fanconi anemia confirmed by a positive test for increased chromosomal breakage with mitomycin C or diepoxybutane from peripheral blood, bone marrow or amniotic fluid.
2. Bone marrow biopsy/aspirate with cellularity (mononuclear cells per ml of bone marrow obtained), CD34+ content (% of MNC), and normal cytogenetics within three months of collection.
3. For the first two cohorts: Absolute neutrophil count > 750/mm3, Hemoglobin > 8 gm/dl without transfusion, platelet count > 50,000/mm3 without transfusion (within 30 days prior to bone marrow collection or PB stem cell mobilization). For the final cohort, the platelet count will be >30,000/mm3 without transfusion (within 30 days prior to bone marrow collection or PB stem cell mobilization).
4. Minimum weight: 7.5 kg.
5. Age:

   First cohort - > 7 Second cohort - > 3 Third cohort - >1.
6. Ability of patient or parent/legal guardian to consent for bone marrow harvest.
7. Ability of patient or parent/legal guardian to consent for placement of temporary apheresis catheter.
8. Ability of patient or parent/legal guardian to consent for apheresis collection.
9. Ability of patient or parent/legal guardian to consent for PRBC/platelet transfusions.

Exclusion Criteria:

1. Myeloid or lymphoid leukemia.
2. Clonal cytogenetic abnormality of bone marrow or peripheral blood lymphocytes (in >2 metaphases by G-banded karyotype or any chromosome deletions of chromosome 7 by Fluorescence in situ hybridization or FISH).
3. Pregnancy or lactation. Women with childbearing potential who are to be collected will be advised that the marrow harvest procedure or the risk of G-CSF used for stem cell mobilization may be teratogenic and will be required to take adequate measures to prevent contraception.
4. Concurrent enrollment in any study using an investigational drug (defined as a drug not approved by the FDA) with the exception of androgens or thyroxine.
5. Physical or emotional status that would prevent compliance, ability to understand treatment plan or adequate follow-up.
6. HIV positive patients.
7. Patients with neoplastic or non-neoplastic disease of any major organ system that would compromise their ability to withstand the bone marrow harvest or apheresis procedure.
8. Patients with uncontrolled (culture or biopsy positive) infection requiring intravenous antivirals, antibiotics, or antifungals. Patients on prolonged antifungal therapy are still eligible if they are culture or biopsy negative in residual radiographic lesions, and they meet the other organ function criteria.
9. Patients unable to tolerate general anesthesia.
10. Known adverse reaction to E. coli products or G-CSF and any contraindication to leukocytosis or hypocalcemia or (where indicated) central line placement.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stella Davies, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AMD3100
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AMD3100
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Safely Received AMD3100 Used in Combination With Standard Dose G-CSF
Description: The safety of AMD3100 used in combination with standard dose G-CSF in Fanconi anemia patients to mobilize peripheral blood CD34+ cells for peripheral blood apheresis.
Time Frame: 30 days
Population: Please refer to the adverse event tables for specifics.
Measure: Number; unit: participants
Arm/Group | AMD3100
Number analyzed (Participants) | 1
participants | 1

2. Primary Outcome: Number of Participants for Whom a Sufficient Number of CD34+ Cells Were Mobilized Into the Peripheral Blood
Description: The effectiveness of AMD3100 used in combination with standard dose G-CSF in Fanconi anemia patients to mobilize a sufficient number of CD34+ cells into the peripheral blood. This target number is defined as > 5 CD34+ cells/mm3.
Time Frame: 3 days
Measure: Number; unit: participants
Arm/Group | AMD3100
Number analyzed (Participants) | 1
participants | 1

3. Secondary Outcome: Number of Participants for Whom the Target Number of Hematopoietic Cells Were Collected by Peripheral Blood Apheresis
Description: Collecting a sufficient number of hematopoietic cells by peripheral blood apheresis, in patients with Fanconi anemia mobilized by AMD3100/G-CSF. This target number is defined as 2 x 106 CD34+ cells per kg patient weight based on the predicted weight in 5 years.
Time Frame: 3 days
Measure: Number; unit: participants
Arm/Group | AMD3100
Number analyzed (Participants) | 1
participants | 1

4. Secondary Outcome: Number of Participants for Whom the Target Number of CD34+ Cells Were Collected From Their Bone Marrow
Description: To collect a sufficient number of CD34+ cells from the bone marrow of Fanconi anemia patients who have failed AMD3100/G-CSF mobilization. This target number is defined as 2 x 106 CD34+ cells per kg patient weight based on the predicted weight in 5 years.
Time Frame: 3 days
Population: One patient was enrolled and this patient met the target for collection.
Measure: Number; unit: participants
Arm/Group | AMD3100
Number analyzed (Participants) | 1
participants | 1

5. Secondary Outcome: Number of Participants for Whom the Target Number of CD34+ Cells Were Isolated.
Description: Isolating a sufficient number of CD34+ cells for clinical studies using the AmCell CliniMACs selection system. This target number is defined as 1 x 106 CD34+ cells per kg patient weight based on the predicted weight in 5 years.
Time Frame: 3 days
Measure: Number; unit: participants
Arm/Group | AMD3100
Number analyzed (Participants) | 1
participants | 1

6. Secondary Outcome: Number of Participants Whose Product Was Used for Preclinical Biological Investigations.
Description: To provide cells for preclinical biological investigations (up to 10% of the final product may be used).
Time Frame: 3 days
Measure: Number; unit: participants
Arm/Group | AMD3100
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Time Frame: 30 days following the last dose of AMD3100
Arm/Group | AMD3100
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMD3100 (N=1)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3)
Hypotension (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes